CLINICAL TRIAL: NCT01471171
Title: A Multiple Dose, Randomised, Double-blind, Placebo Controlled, 2 Period Crossover Clinical Trial to Assess the Effect of Aclidinium Bromide 400 μg BID on Exercise Endurance in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Aclidinium Bromide 400 µg BID (Twice a Day)Compared to Placebo in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/40
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Antimuscarinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium bromide (Experimental): 3-week treatment periods
  Interventions: Drug: Aclidinium Bromide
- Placebo (Experimental): 3-week treatment periods
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium Bromide — 1 puff of 400 micro grams in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h)
  Arms: Aclidinium bromide
Drug: Placebo — 1 puff of placebo in the morning (09:00 ± 1h) and 1 puff in the evening (21:00 ± 1h)
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the effect of aclidinium bromide 400 μg twice a day (BID) administered twice a day versus placebo on exercise endurance and on hyperinflation and dyspnoea at rest and during exercise after 3 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients aged ≥ 40 with stable moderate to severe COPD (Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines).
* Post-salbutamol Forced Expiratory Volume in one second(FEV1) < 80% and ≥ 30% of predicted normal value and Post-salbutamol FEV1/Forced Vital Capacity (FVC) < 70%.
* Current or ex-smokers of ≥ 10 pack-years
* Functional residual capacity (FRC) measured by body plethysmography at Screening Visit ≥ 120% of predicted value

Exclusion Criteria:

* History or current diagnosis of asthma
* Signs of an exacerbation within 6 weeks ( or 3 months if results in hospitalisation) prior to the screening visit or during the run-in period.
* Clinically significant respiratory and/or cardiovascular conditions or laboratory abnormalities.
* Conditions where the use of anticholinergic drugs is contraindicated, such as known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma.
* Patients with an oxygen saturation < 85% during cycle exercise on room air at Screening Visit, Run- in Visit and Visit 1.
* Contra-indications of cardiopulmonary exercise testing.
* Patient who in the investigator's opinion will need to start a pulmonary rehabilitation program during the study and/or patients who have just started/finished pulmonary rehabilitation at least 3 months prior to the Screening Visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, Ph.D., Study Director — AstraZeneca
Locations (14):
- Germany (10):
  - Almirall Investigational Site #10, Berlin
  - Almirall Investigational Site #6, Berlin
  - Almirall Investigational Site #2, Berlin
  - Almirall Investigational Site #4, Frankfurt
  - Almirall Investigational Site #5, Großhansdorf
  - Almirall Investigational Site #8, Hamburg
  - Almirall Investigational Site #9, Hamburg
  - Almirall Investigational Site #3, Hanover
  - Almirall Investigational Site #7, Lübeck
  - Almirall Investigational Site #1, Wiesbaden
- Spain (3):
  - Almirall Investigational Site #1, Alicante
  - Almirall Investigational Site #4, Barcelona
  - Almirall Investigational Site #2, Madrid
- Almirall Investigational Site #2, London, United Kingdom

REFERENCES:
- [Derived] Beeh KM, Watz H, Puente-Maestu L, de Teresa L, Jarreta D, Caracta C, Garcia Gil E, Magnussen H. Aclidinium improves exercise endurance, dyspnea, lung hyperinflation, and physical activity in patients with COPD: a randomized, placebo-controlled, crossover trial. BMC Pulm Med. 2014 Dec 23;14:209. doi: 10.1186/1471-2466-14-209. PMID 25539654
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3974&filename=Synopsis-las40-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 enrolling sites. A total of 14 sites randomised patients: 10 sites in Germany, 3 sites in Spain and one site in the United Kingdom. The first patient was screened in November 2011 and the last patient visit was in June 2012.
Pre-assignment Details: Eligible patients entered a 14-21 day run-in period to assess disease stability. During this period, one site visit was performed to familiarise patients with study testing procedures (body plethysmography, spirometry and a constant work rate cycle exercise test).
Groups:
- Aclidinium Bromide 400 μg - Placebo: The study consisted of 2 treatment periods of 22 (±2) days separated by a washout period of 14 (-2/+7) days. In treatment period 1, patients received 1 puff of aclidinium bromide 400 μg via the Genuair® multidose dry powder inhaler in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h) for 3 weeks. In treatment period 2, patients received 1 puff of placebo via the Genuair® multidose dry powder inhaler in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h) for 3 weeks.
- Placebo - Aclidinium Bromide 400 μg: The study consisted of 2 treatment periods of 22 (±2) days separated by a washout period of 14 (-2/+7) days. In treatment period 1, patients received 1 puff of placebo via the Genuair® multidose dry powder inhaler in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h) for 3 weeks. In treatment period 2, patients received 1 puff of aclidinium bromide 400 μg via the Genuair® multidose dry powder inhaler in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h) for 3 weeks.
Period: Treatment Period 1
Arm/Group | Aclidinium Bromide 400 μg - Placebo | Placebo - Aclidinium Bromide 400 μg
Started | 57 | 55
Completed | 53 | 54
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 1
Period: Treatment Period 2
Arm/Group | Aclidinium Bromide 400 μg - Placebo | Placebo - Aclidinium Bromide 400 μg
Started | 53 | 54
Completed | 52 | 54
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Safety Population: All patients randomized into the crossover study were included in the safety population
Arm/Group | Overall Study Safety Population
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.1)
Gender [Count of Participants; unit: Participants]
  Female | 36
  Male | 76
Region of Enrollment [Number; unit: participants]
  Spain | 20
  Germany | 89
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endurance Time (Seconds)
Description: Change from baseline in endurance time during constant work rate cycle ergometry to symptom limitation at 75% of Maximum Work load (Wmax) after 3 weeks of treatment.
Time Frame: Week 3
Population: Intention-to-Treat (ITT) population: all randomised patients who took at least one dose of investigational medicinal product, and had at least a baseline and one post-dose corresponding assessment value of the primary efficacy variable in one of the 2 treatment periods. 2 patients from the safety population were excluded from the ITT population.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Groups:
- Aclidinium Bromide 400 μg Bid: Aclidinium bromide: Oral inhalation via Genuair® multidose dry powder inhaler. 1 puff of 400 μg in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h) for 3 weeks.
- Placebo: Placebo: Oral inhalation by Genuair® multidose dry powder inhaler. 1 puff of placebo in the morning (09:00 ± 1h) and 1 puff in the evening (21:00 ± 1h) for 3 weeks.
Arm/Group | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 109 | 107
Seconds | 68.3 (18.8) | 9.8 (19.0)

2. Secondary Outcome: Change From Baseline in Trough Inspiratory Capacity (IC) (Litres)
Description: Change from baseline in trough IC after 3 weeks of treatment
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 107 | 104
Litres | 0.098 (0.024) | 0.020 (0.025)

3. Secondary Outcome: Change From Baseline in Intensity of Dyspnoea
Description: Change from baseline in intensity of dyspnoea based on the Borg CR10 Scale® (ranging from '0'=nothing at all to '10'=extremely strong/maximal dyspnoea, the highest possible numerical value) at isotime during constant work rate cycle ergometry after 3 weeks of treatment.
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 109 | 107
Units on a scale | -0.48 (0.20) | 0.15 (0.20)

ADVERSE EVENTS:
Arm/Group | Aclidinium Bromide 400 μg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/111 | 2/108
Other Adverse Events (participants affected / at risk) | 7/111 | 4/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 400 μg Bid (N=111) | Placebo (N=108)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Preferred term was coded as chronic obstructive pulmonary disease (COPD). However, per protocol, only COPD exacerbations (worsening of COPD symptoms for at least 2 consecutive days that required a change in COPD treatment) were reported as AEs.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 400 μg Bid (N=111) | Placebo (N=108)
Nasopharyngitis (Infections and infestations) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.